CLINICAL TRIAL: NCT07061067
Title: Affection of Symptoms Duration on Outcomes of Lumbar Spine Surgery
Status: Recruiting | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ayman Mohamed Basha, Lecturer of Neurosurgery, Faculty of Medicine, KafrElsheikh University, KafrElsheikh, Egypt, Kafrelsheikh University
Other Study IDs: KFSIRB200-644
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Symptom Duration; Outcomes; Lumbar Spine Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients undergoing lumbar spine surgery
  Interventions: Procedure: Lumbar Spine Surgery

INTERVENTIONS:
Procedure: Lumbar Spine Surgery — Patients undergoing lumbar spine surgery Presenting symptoms include lumbar back pain, lumbar radiculopathy, neurogenic claudication, lower-extremity weakness, bowel or bladder symptoms, and duration of symptoms.

SUMMARY:
This study aims to evaluate the affection of symptoms duration on outcomes of lumbar spine surgery.

DETAILED DESCRIPTION:
Lumbar spine surgery is a pivotal intervention for a variety of conditions affecting the lower back, such as degenerative disc disease, spinal stenosis, spondylolisthesis, and disc herniation.

The first line of treatment in lumbar spine is usually conservative. If conservative treatment fails to lead to an improvement in symptoms in 3 to 6 months, surgical treatment can be considered as an option for symptom relief. Invasive therapies are considered when neurogenic claudication is present with positive findings from diagnostic imaging. Surgery has been shown to provide better outcomes for at least 4 years in terms of disability and pain with a narrowing of the benefits over time compared with conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Both sexes.
* Patients undergoing lumbar spine surgery
* Presenting symptoms include lumbar back pain, lumbar radiculopathy, neurogenic claudication, lower-extremity weakness, bowel or bladder symptoms, and duration of symptoms.

Exclusion Criteria:

* Previous spinal surgery.
* Vascular claudication.
* Comorbid pathology affecting walking ability.
* Severe comorbidities that may impact surgery outcomes (e.g., uncontrolled diabetes, cardiovascular disease).
* Bony metastases.
* Unfit for general anaesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study will be carried out on 60 patients undergoing lumbar spine surgery admitted in KafrElsheikh University Hospitals over a period of 6 months starting from approval of the Medical Sciences Ethics Committee of KafrElsheikh Faculty of Medicine and all the included patients will provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-19 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Disability assessment | 6 months postoperatively
  Disability assessment will be done by the Oswestry Disability Index (ODI). ODI is a pain-related disability score ranging from 0 (no impairment) to 100 (bedbound).

SECONDARY OUTCOMES:
Degree of pain | 6 months postoperatively
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable").
Musculoskeletal conditions | 6 months postoperatively
  Global Perceived Effect (GPE) will be used to assess musculoskeletal conditions like neck pain. The GPE scale has seven steps (1=completely recovered, 2=much improved, 3=somewhat improved, 4=unchanged, 5=somewhat worse, 6=much worse, 7=worse than ever)
Degree of patient satisfaction | 6 months postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.